CLINICAL TRIAL: NCT01909466
Title: An Open-label, Multiple Dose, Safety and Tolerability Study of Aripiprazole IM Depot Administered in the Deltoid Muscle in Adult Subjects With Schizophrenia
Brief Title: Safety and Tolerability Study of Aripiprazole IM Depot in Adult Subjects With Schizophrenia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 31-12-298
Record Dates: First submitted 2013-07-24; First posted 2013-07-26 (Estimated); Results first posted 2015-06-02 (Estimated); Last update posted 2015-07-01 (Estimated); Status verified 2015-06

CONDITIONS: Schizophrenia; Mental Disorder; Nervous System Diseases
Keywords: OPC-14597; Aripiprazole; Schizophrenia
MeSH Terms: conditions — Schizophrenia; Mental Disorders; Nervous System Diseases | interventions — Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gluteal Injection (Other)
  Interventions: Drug: Aripiprazole, OPC-14597
- Deltoid Injection (Other)
  Interventions: Drug: Aripiprazole, OPC-14597

INTERVENTIONS:
Drug: Aripiprazole, OPC-14597 — 5 monthly applications of 400 mg of aripiprazole IM depot, where the first application is in the gluteal or deltoid muscle followed by 4 monthly administrations to the deltoid muscle

SUMMARY:
To determine the safety and tolerability of multiple-dose administrations of aripiprazole intramuscular (IM) depot in the deltoid muscle in adult subjects with schizophrenia

DETAILED DESCRIPTION:
This is a trial designed to assess the safety and tolerability of multiple-dose administrations of aripiprazole intramuscular (IM) depot in the deltoid muscle in adult subjects with schizophrenia. The trial consists of a 113 day treatment period with a 28 day followup. The trial population will include male and female subjects between 18 and 64 years (inclusive), with a current diagnosis of schizophrenia as defined by DSM-IV-TR criteria and a prior history of tolerating aripiprazole per investigator's judgement.

ELIGIBILITY:
Inclusion Criteria:

* Male and female individuals between 18 and 64 years, inclusive, at the time of informed consent.
* Prior history of tolerating aripiprazole per investigator's judgement.

Exclusion Criteria:

* Subjects who have met DSMV-IV-TR criteria for substance dependence within the past 180 days.
* Subjects who use more than one antipsychotic medication at screening.
* Use of any CYP2D6 and CYP3A4 inhibitors, or CYP3A4 inducers within 14 days prior to dosing and for the duration of the trial.
* Subjects who participated in any clinical trial involving a psychotropic medication within 1 month prior to enrollment.
* Subjects currently in an acute relapse of schizophrenia.
* Subjects with a current DSMV-IV-TR diagnosis other than schizophrenia.
* Subjects who are considered treatment-resistant to antipsychotic medications.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 141 (Actual)
Dates: Start 2013-07; Primary Completion 2014-03 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Largay, MD, Study Director — Otsuka Pharmaceutical Development & Commercialization, Inc.
Locations (11):
- United States (11):
  - Comprehensive Clinical Development, Cerritos, California
  - Collaborative Neuroscience Network, Inc., Garden Grove, California
  - CNRI-San Diego, San Diego, California
  - Comprehensive Clinical Development, Washington D.C., District of Columbia
  - Scientific Clinical Research, Inc., Fort Lauderdale, Florida
  - Compass Research North, LLC, Leesburg, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - St. Louis Clinical Trials, St Louis, Missouri
  - CRI Lifetree, Marlton, New Jersey
  - CRI Lifetree, Philadelphia, Pennsylvania
  - Community Clinical Research, Inc., Austin, Texas

REFERENCES:
- [Derived] Raoufinia A, Peters-Strickland T, Nylander AG, Baker RA, Eramo A, Jin N, Bricmont P, Repella J, McQuade RD, Hertel P, Larsen F. Aripiprazole Once-Monthly 400 mg: Comparison of Pharmacokinetics, Tolerability, and Safety of Deltoid Versus Gluteal Administration. Int J Neuropsychopharmacol. 2017 Apr 1;20(4):295-304. doi: 10.1093/ijnp/pyw116. PMID 28204607

RESULTS

PARTICIPANT FLOW:
Recruitment Details: An open-label, multiple dose, multiple-site trial of adult participants with schizophrenia for the first application of aripiprazole intramuscular (IM) depot 400 mg in the gluteal or deltoid muscle (1:1 ratio) followed by 4 monthly administrations to the deltoid muscle site in all participants.
Pre-assignment Details: Prior to the trial, the participants were stabilized for at least 14 days on their current oral antipsychotic medication prior to administration of the first aripiprazole IM depot.
Groups:
- Gluteal/Deltoid: Participants were injected with aripiprazole IM depot 400 mg at the gluteal muscle site on Day 1 and followed by 4 subsequent deltoid administrations every 28 days.
- Deltoid/Deltoid: Participants were injected with aripiprazole IM depot 400 mg at the deltoid muscle site on Day 1 and followed by 4 subsequent deltoid administrations every 28 days.
Period: Overall Study
Arm/Group | Gluteal/Deltoid | Deltoid/Deltoid
Started | 68 | 73
Completed | 46 | 50
Not Completed | 22 | 23
Not completed — Lost to Follow-up | 5 | 7
Not completed — Adverse Event | 3 | 4
Not completed — Met Withdrawal Criteria | 0 | 3
Not completed — Physician Decision | 2 | 0
Not completed — Withdrawal by Subject | 11 | 9
Not completed — Lack of Efficacy | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Aripiprazole IM Depot 400 mg - Total: Participants were injected with aripiprazole IM depot 400 mg at the deltoid/ gluteal muscle site on Day 1 and followed by 4 subsequent deltoid administrations every 28 days.
Arm/Group | Aripiprazole IM Depot 400 mg - Total
Number analyzed (Participants) | 141
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.9 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 109

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs).
Description: AE was defined as any new medical problem, or exacerbation of an existing problem, experienced by a participant while enrolled in the trial, whether or not it was considered drug related by the investigator. A serious adverse event (SAE) was any untoward medical occurrence that resulted in death or was life threatening or required inpatient hospitalization or prolonged hospitalization. A treatment-emergent AE (TEAE) was defined as an AE that started after start of study medication or an AE that continued from baseline and that worsened, was serious, was study medication related, or resulted in death, discontinuation, interruption, or reduction of study medication.
Time Frame: AEs were recorded from the time the informed consent was signed until follow-up for 28 days after last
Population: The safety sample included all randomized participants who were administered at least one dose of study medication, regardless of any protocol violation.
Measure: Number; unit: participants
Arm/Group | Aripiprazole IM Depot 400 mg - Total
Number analyzed (Participants) | 138
participants
  Participants with TEAEs | 112
  Participants with serious TEAEs | 4
  Participants with non-serious TEAEs | 112
  Participants with severe TEAEs | 2

2. Primary Outcome: Mean Visual Analog Scale (VAS) Score for Rating of Pain at the Injection Site.
Description: Participants assessed the pain associated with injection of aripiprazole IM using the VAS instrument. This was done approximately 30 minutes pre-dose and 1 hour (±15 min) Post-dose on Days 1, 29, 57, 85 and 113. For the first injection, the pre-dose assessment was of the current injection site. For the injections 2 through 5, the pre-dose assessment was of the prior injection site. Investigator's Assessment of Most Recent Injection Site including pain, swelling, redness, and induration were reported in 4-point categorical scale (1 = absent, 2 = mild, 3 = moderate and 4 = severe) by first injection site at each injection.
Time Frame: Days 1 and 113
Population: The safety sample included all randomized participants who were administered at least one dose of study medication, regardless of any protocol violation. In LOCF dataset, missing data at a post-baseline visit were imputed with the value obtained at the nearest preceding visit.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Aripiprazole IM Depot 400 mg - Total
Number analyzed (Participants) | 138
Units on a scale
  First injection (Day 1) | 2.0 (4.4)
  Last injection (Day 113) | 1.2 (3.4)

3. Primary Outcome: Mean Change From Baseline in Suicidal Ideation Intensity Total Score Via Columbia-suicide Severity Rating Scale (C-SSRS).
Description: Suicidality was monitored throughout the trial using C-SSRS. The C-SSRS addresses the need for standardized classification of suicide reports to assess suicide risk. This scale consisted of Baseline evaluation that assessed the lifetime experience of the participant with suicidal events and suicidal ideation and a post baseline evaluation that focuses on suicidality since the last trial visit. The C-SSRS since last visit form were completed on Day 1 pre-dose and prior to dosing on Days 29, 57, 85, 113, 141/ Early Termination(ET) and prior to pharmacokinetics(PK) sampling on Days 8, 15, 22, 120, 127 and 134. The suicidal ideation intensity total score was the sum of suicidal ideation severity rating scores for frequency, duration, controllability, deterrents, and reasons for ideation. For each item, each participant got an intensity score from 0(none) to 5(worst). Therefore,the suicidal ideation intensity total score range from 0 to 25, with a score of 0 given for no suicidal ideation.
Time Frame: Baseline to Last Visit (Day 141)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Aripiprazole IM Depot 400 mg - Total
Number analyzed (Participants) | 138
Units on a scale
  Week 1 (N= 135) | 0.0 (0.0)
  Week 2 (N= 132) | 0.0 (0.0)
  Week 3 (N= 131) | 0.0 (0.0)
  Week 4 (N= 129) | 0.2 (1.3)
  Week 8 (N= 112) | 0.1 (1.0)
  Week 12 (N= 109) | 0.1 (1.1)
  Week 16 (N= 99) | 0.0 (0.0)
  Week 17 (N=100) | 0.0 (0.0)
  Week 18 (N= 98) | 0.0 (0.0)
  Week 19 (N= 99) | 0.0 (0.0)
  Week 20 (N= 97) | 0.0 (0.0)
  Last Visit (N= 136) | 0.1 (0.6)

4. Primary Outcome: Mean Change From Baseline Measured by Extrapyramidal Symptoms (EPS) by Simpson-Angus Scale (SAS).
Description: The SAS consisted of a list of 10 symptoms of Parkinsonism (gait, arm dropping, shoulder shaking, elbow rigidity, wrist rigidity, head rotation, glabella tap, tremor, salivation, and akathisia). The SAS Total Score was the sum of the scores for all 10 items. SAS total score can range from 10 to 50. Each item was rated on a 5-point scale, with a score of 1 =absence of symptoms and a score of 5 =severe condition.
Time Frame: Baseline to Week 20
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Aripiprazole IM Depot 400 mg - Total
Number analyzed (Participants) | 138
Units on a scale
  Week 1(N= 135) | 0.01 (0.89)
  Week 2 (N= 136) | 0.04 (0.83)
  Week 3 (N= 136) | -0.02 (1.08)
  Week 4 (N= 136) | 0.01 (0.98)
  Week 8 (N= 136) | 0.02 (1.11)
  Week 12 (N= 136) | 0.04 (1.17)
  Week 16 (N= 136) | 0.07 (1.04)
  Week 20 (N= 136) | 0.07 (1.20)

5. Primary Outcome: Mean Change From Baseline Measured by EPS by Abnormal Involuntary Movement Scale (AIMS).
Description: The AIMS assessment consisted of 10 items describing symptoms of dyskinesia. Facial and oral movements (items 1 through 4), extremity movements (items 5 and 6), and trunk movements (item 7) were observed unobtrusively while the participant was at rest (e.g., in the waiting room), and the study physician would make global judgments on the participant's dyskinesia's (items 8 through 10). These items are rated on a five-point scale of severity from 0-4. The scale is rated from 0 (none), 1 (minimal), 2 (mild), 3 (moderate), 4 (severe). Overall AIMS scores range from 0 to 42.
Time Frame: Baseline to Week 20
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Aripiprazole IM Depot 400 mg - Total
Number analyzed (Participants) | 138
Units on a scale
  Week 1(N= 135) | -0.03 (0.42)
  Week 2 (N= 136) | -0.05 (0.37)
  Week 3 (N= 136) | -0.01 (0.52)
  Week 4 (N= 136) | -0.03 (0.50)
  Week 8 (N= 136) | -0.05 (0.53)
  Week 12 (N= 136) | 0.00 (0.40)
  Week 16 (N= 136) | -0.03 (0.52)
  Week 20 (N= 136) | 0.03 (0.64)

6. Primary Outcome: Mean Change From Baseline Measured by EPS by Barnes Akathisia Rating Scale (BARS).
Description: The BARS consisted of 4 items related to akathisia: objective observation of akathisia by the study physician, subjective feelings of restlessness by the participant, participant distress due to akathisia, and global evaluation of akathisia. To complete this scale, participants were observed while they were seated and then stood for a minimum of 2 minutes in each position. Symptoms observed in other situations (e.g., while engaged in neutral conversation or engaged in activity on the ward) may also be rated. Subjective phenomena were to be elicited by direct questioning. The first 3 items were rated on a 4-point scale, with a score of 0 = absence of symptoms and a score of 3 = severe condition. The global clinical evaluation were made on a 6-point scale, (0=absent, 1=questionable, 2=mild, 3=moderate, 4=marked, 5=severe).
Time Frame: Baseline to Week 20
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Aripiprazole IM Depot 400 mg - Total
Number analyzed (Participants) | 138
Units on a scale
  Week 1(N=135) | 0.03 (0.47)
  Week 2 (N=136) | 0.08 (0.50)
  Week 3 (N=136) | 0.08 (0.57)
  Week 4 (N=136) | 0.06 (0.47)
  Week 8 (N=136) | 0.11 (0.59)
  Week 12 (N=136) | 0.06 (0.51)
  Week 16 (N=136) | 0.06 (0.51)
  Week 20 (N=136) | 0.04 (0.47)

7. Secondary Outcome: Mean Change From Baseline in Total Score of Positive and Negative Syndrome Scale (PANSS).
Description: The PANSS consisted of three subscales: a total of 30 symptom constructs. For each symptom construct, severity was rated on a 7-point scale, with a score of 1 (absence of symptoms) and a score of 7 (extremely severe symptoms). The PANSS total score was the sum of the rating scores for 7 positive scale items, 7 negative scale items, and 16 general psychopathology scale items from the PANSS panel. The PANSS total score ranged from 30 (best possible outcome) to 210 (worst possible outcome).
Time Frame: Baseline to Week 20
Population: In efficacy analysis, the dataset included all randomized participants who received at least one dose of aripiprazole IM depot injection and had at least one efficacy assessment. In LOCF dataset, missing data at a post-baseline visit were imputed with the value obtained at the nearest preceding visit.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Aripiprazole IM Depot 400 mg - Total
Number analyzed (Participants) | 138
Units on a scale
  Week 8 (N= 128) | -0.94 (9.42)
  Week 20 (N= 128) | -2.23 (10.95)

8. Secondary Outcome: Mean Change From Baseline in PANSS Positive Sub-scale Score.
Description: The PANSS consisted of three subscales: a total of 30 symptom constructs. For each symptom construct, severity was rated on a 7-point scale, with a score of 1 (absence of symptoms) and a score of 7 (extremely severe symptoms). The PANSS positive subscale score was the sum of the rating scores for the 7 positive scale items from the PANSS panel. The 7 positive symptom constructs are delusions, conceptual disorganization, hallucinatory behavior, excitement, grandiosity, suspiciousness/persecution, and hostility. The PANSS Positive Subscale ranges from 7 (absence of symptoms) to 49 (extremely severe symptoms).
Time Frame: Baseline to Week 20
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Aripiprazole IM Depot 400 mg - Total
Number analyzed (Participants) | 138
Units on a scale
  Week 8 (N= 128) | -0.14 (3.18)
  Week 20 (N= 128) | -0.52 (3.84)

9. Secondary Outcome: Mean Change From Baseline in PANSS Negative Sub-scale Score.
Description: The PANSS consisted of three subscales: a total of 30 symptom constructs. For each symptom construct, severity was rated on a 7-point scale, with a score of 1 (absence of symptoms) and a score of 7 (extremely severe symptoms). The PANSS negative subscale score was the sum of the rating scores for the 7 negative scale items from the PANSS panel. The 7 negative symptom constructs: blunted affect, emotional withdrawal, poor rapport, passive apathetic withdrawal, difficulty in abstract thinking, lack of spontaneity and flow of conversation, stereotyped thinking. The PANSS Negative Subscale ranges from 7 (absence of symptoms) to 49 (extremely severe symptoms).
Time Frame: Baseline to Week 20
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Aripiprazole IM Depot 400 mg - Total
Number analyzed (Participants) | 138
Units on a scale
  Week 8 (N= 128) | -0.30 (3.56)
  Week 20 (N= 128) | -0.33 (3.79)

10. Secondary Outcome: Mean Change From Baseline in Clinical Global Impression-Severity (CGI-S) Score.
Description: The severity of illness for each participant was rated using the CGI-S scale. To assess CGI-S, the study physician answered the following question: "Considering your total clinical experience with this particular population, how mentally ill is the participant at this time?" Response choices included: 0 = not assessed; 1 = normal, not ill at all; 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; and 7 = among the most extremely ill participants.
Time Frame: Baseline to Week 20
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Aripiprazole IM Depot 400 mg - Total
Number analyzed (Participants) | 138
Units on a scale
  Week 8 (N= 128) | -0.02 (0.57)
  Week 20 (N= 128) | -0.09 (0.61)

11. Secondary Outcome: Clinical Global Impression-Improvement (CGI-I) Score.
Description: The efficacy of trial medication were rated for each participant using the CGI-I scale. The study physician must rate the participant's total improvement whether or not it is due entirely to drug treatment. All responses were compared to the participant's condition a baseline. Response choices include: 0 = not assessed; 1 =very much improved; 2 = much improved; 3 = minimally improved; 4 = no change; 5 =minimally worse; 6 = much worse; and 7 = very much worse.
Time Frame: Baseline to Week 20
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Aripiprazole IM Depot 400 mg - Total
Number analyzed (Participants) | 138
Units on a scale
  Week 8 (N= 128) | 3.86 (0.78)
  Week 20 (N= 128) | 3.70 (0.98)

12. Secondary Outcome: Mean Change From Baseline in Total Score of Subject Well-being Under Neuroleptic Treatment-Short Form (SWN-S).
Description: The participant's feeling of their own well-being was assessed using the 20 question SWN-S. The SWN-S was a validated self-report instrument that evaluated the participant's perception of 1 being while receiving antipsychotic medication. The questionnaire consisted of 20 items and 5 subscales (mental functioning, social integration, emotional regulation, physical functioning, self-control) whose items followed in random order. For items marked with a '+', response choices and scoring were as follows: not at all = 1, hardly at all = 2, a little = 3, somewhat = 4, much = 5, very much = 6. For items marked with a '-', the scoring was reversed; response choices and scoring were as follows: not at all = 6, hardly at all = 5, a little = 4, somewhat = 3, much = 2, very much = 1. The total score from the scale ranges from 20 (bad subjective experience) to 120 (perfect subjective experience).
Time Frame: Baseline to Week 20+
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Aripiprazole IM Depot 400 mg - Total
Number analyzed (Participants) | 138
Units on a scale
  Week 8 (N= 128) | -1.17 (15.95)
  Week 20 (N= 128) | -0.81 (17.09)

13. Secondary Outcome: Mean Change From Baseline in Mental Functioning Score of SWN-S.
Description: The participant's feeling of their own well-being was assessed using the 20 question SWN-S. The SWN-S was a validated self-report instrument that evaluated the participant's perception of 1 being while receiving antipsychotic medication. The questionnaire consisted of 20 items and 5 subscales (mental functioning, social integration, emotional regulation, physical functioning, self-control) whose items followed in random order. For items marked with a '+', response choices and scoring were as follows: not at all = 1, hardly at all = 2, a little = 3, somewhat = 4, much = 5, very much = 6. For items marked with a '-', the scoring was reversed; response choices and scoring were as follows: not at all = 6, hardly at all = 5, a little = 4, somewhat = 3, much = 2, very much = 1. SWN-S subscale score's each item was rated on a score of 0 (none) to 6 (severe), with higher scores indicating stronger subjective feelings of deficit.
Time Frame: Baseline to Week 20
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Aripiprazole IM Depot 400 mg - Total
Number analyzed (Participants) | 138
Units on a scale
  Week 8 (N= 128) | -0.18 (4.85)
  Week 20 (N= 128) | 0.01 (4.83)

14. Secondary Outcome: Mean Change From Baseline in Self Control Score of SWN-S.
Description: as for outcome 13
Time Frame: Baseline to Week 20
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Aripiprazole IM Depot 400 mg - Total
Number analyzed (Participants) | 138
Units on a scale
  Week 8 (N= 128) | -0.47 (3.90)
  Week 20 (N= 128) | -0.64 (4.14)

15. Secondary Outcome: Mean Change From Baseline in Physical Functioning Score of SWN-S.
Description: as for outcome 13
Time Frame: Baseline to Week 20
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Aripiprazole IM Depot 400 mg - Total
Number analyzed (Participants) | 138
Units on a scale
  Week 8 (N= 128) | -0.39 (4.44)
  Week 20 (N= 128) | -0.37 (4.34)

16. Secondary Outcome: Mean Change From Baseline in Emotional Regulation Score of SWN-S.
Description: as for outcome 13
Time Frame: Baseline to Week 20
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Aripiprazole IM Depot 400 mg - Total
Number analyzed (Participants) | 138
Units on a scale
  Week 8 (N= 128) | 0.30 (3.36)
  Week 20 (N= 128) | 0.46 (4.05)

17. Secondary Outcome: Mean Change From Baseline in Social Integration Score of SWN-S.
Description: as for outcome 13
Time Frame: Baseline to Week 20
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Aripiprazole IM Depot 400 mg - Total
Number analyzed (Participants) | 138
Units on a scale
  Week 8 (N= 128) | -0.47 (4.28)
  Week 20 (N= 128) | -0.32 (4.43)

ADVERSE EVENTS:
Time Frame: Adverse events were reported from the signing of the ICF until follow-up for up to 28 days after the last dose of study medication.
Description: A SAE was an untoward medical occurrence resulted in death or required inpatient hospitalization or prolonged hospitalization. An AE was an exacerbation of an existing problem or a new problem experienced by a participant when enrolled in a trial whether or not it was considered drug related by study physician.
Arm/Group | Aripiprazole IM Depot 400 mg - Total
Serious Adverse Events (participants affected / at risk) | 4/138
Other Adverse Events (participants affected / at risk) | 112/138
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aripiprazole IM Depot 400 mg - Total (N=138)
Atrial fibrillation (Cardiac disorders) | 1
Psychotic disorder (Psychiatric disorders) | 1
Schizophrenia (Psychiatric disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aripiprazole IM Depot 400 mg - Total (N=138)
Diarrhoea (Gastrointestinal disorders) | 7
Dyspepsia (Gastrointestinal disorders) | 9
Nausea (Gastrointestinal disorders) | 9
Toothache (Gastrointestinal disorders) | 11
Injection site pain (General disorders) | 38
Upper respiratory tract infection (Infections and infestations) | 11
Weight increased (Investigations) | 17
Akathisia (Nervous system disorders) | 11
Headache (Nervous system disorders) | 16
Insomnia (Psychiatric disorders) | 7
Restlessness (Psychiatric disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No